CLINICAL TRIAL: NCT02914275
Title: A Phase 3, Randomized, Multicenter, Observer-blinded, Noninferiority Study to Evaluate the Immunogenicity and Safety of a Quadrivalent Inactivated Influenza Virus Vaccine (Seqirus QIV) With a US-licensed Quadrivalent Inactivated Comparator Influenza Virus Vaccine (Comparator QIV) in a Pediatric Population 6 Months Through 59 Months of Age
Brief Title: A Study to Evaluate the Immunogenicity and Safety of Seqirus Quadrivalent Influenza Vaccine (QIV) in a Pediatric Population 6 Months Through 59 Months of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-QIV-15-03
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2018-11

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Seqirus QIV Cohort A (Experimental): Seqirus Quadrivalent Inactivated Influenza Vaccine - Subjects 6 months through 35 months of age
  Interventions: Biological: Seqirus Quadrivalent Inactivated Influenza Vaccine
- Seqirus QIV Cohort B (Experimental): Seqirus Quadrivalent Inactivated Influenza Vaccine - Subjects 36 months through 59 months of age
  Interventions: Biological: Seqirus Quadrivalent Inactivated Influenza Vaccine
- Comparator QIV Cohort A (Active Comparator): Comparator Quadrivalent Inactivated Influenza Vaccine - Subjects 6 months through 35 months of age
  Interventions: Biological: Comparator Quadrivalent Inactivated Influenza Vaccine
- Comparator QIV Cohort B (Active Comparator): Comparator Quadrivalent Inactivated Influenza Vaccine - Subjects 36 months through 59 months of age
  Interventions: Biological: Comparator Quadrivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: Seqirus Quadrivalent Inactivated Influenza Vaccine — The Seqirus study vaccine is a sterile, thimerosal-free suspension containing 60 mcg total hemagglutinin antigen per 0.5 mL (15 mcg each of the four recommended influenza strains for the Northern Hemisphere 2016/2017 influenza season). Subjects will receive one or two doses according to the recommendations of the Advisory Committee on Immunization Practices for the United States 2016-17 Influenza Season. Preferred sites for intramuscular injection are the anterolateral aspect of the thigh in infants 6 months through 11 months of age, the anterolateral aspect of the thigh (or the deltoid muscle of the arm if muscle mass is adequate) in children 12 months through 35 months of age.
  Other Names: Seqirus QIV
  Arms: Seqirus QIV Cohort A; Seqirus QIV Cohort B
Biological: Comparator Quadrivalent Inactivated Influenza Vaccine — The comparator Quadrivalent Inactivated Influenza vaccine is a US-licensed product containing four recommended influenza strains for the Northern Hemisphere 2016/2017 influenza season. Subjects will receive one or two doses according to the recommendations of the Advisory Committee on Immunization Practices for the United States 2016-17 Influenza Season. Preferred sites for intramuscular injection of the non-dominant arm in children 36 months through 59 months of age.
  Other Names: Comparator QIV
  Arms: Comparator QIV Cohort A; Comparator QIV Cohort B

SUMMARY:
This is a study to assess the immune (antibody) response and safety of a Seqirus split virion, inactivated Quadrivalent Influenza Vaccine (Seqirus QIV), in comparison with a US licensed 2016/2017 Quadrivalent Influenza Vaccine (comparator QIV) in a healthy pediatric population 6 months through 59 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject 6 months through to 59 months of age at the time of first vaccination and born between 36 and 42 weeks of gestation;
* Parent or legally acceptable representative able to provide written informed consent and be willing and able to adhere to all protocol requirements including blood draws.
* Subject is in generally good health as per the Investigator's medical judgment

Exclusion Criteria:

* History of allergic reactions to egg proteins or any components of the Study Vaccines;
* History of serious adverse reactions to any influenza vaccines;
* History of Guillain-Barré syndrome or other demyelinating disease such as encephalomyelitis and transverse myelitis;
* History of licensed or investigational influenza vaccination in the last 6 months;
* Clinical signs of active infection and/or an axillary temperature of ≥ 99.5°F / (≥ 37.5 °C) on the day of vaccination or within 48 hours preceding vaccination.
* Current or recent, acute or chronic medical conditions that in the opinion of the Investigator are clinically significant and/or unstable
* History of any seizures, with the exception of a single febrile seizure;
* Self-reported or known seropositivity suggestive of acute or chronic viral infection for human immunodeficiency virus, hepatitis B or hepatitis C;
* Known or suspected congenital or acquired immunosuppressive conditions;
* Current or recent immunosuppressive or immunomodulatory therapy
* Current or medical history of malignant neoplasms;
* Administration of immunoglobulin and/or any blood products within the previous 90 days preceding the administration of the Study Vaccine or planned administration during the study;
* Participation in a clinical trial or use of an investigational compound within 28 days prior to or 28 days after receiving the Study Vaccine, or plans to enter a study during this period;
* Vaccination with a licensed vaccine 21 days (for live or inactivated vaccines) prior to receiving the Study Vaccine, or plans to receive any licensed vaccine prior to the Study Exit Visit.
* Medical conditions or treatment contraindicating intramuscular vaccination due to increased risk of bleeding.
* Family members of the employees of the Investigator or study center with direct involvement in the study, or with other clinical studies under the direction of that Investigator or study center.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2250 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-08-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Site 434, Birmingham, Alabama
  - Site 442, Mobile, Alabama
  - Site 430, Anaheim, California
  - Site 437, Anaheim, California
  - Site 423, Downey, California
  - Site 397, Ontario, California
  - Site 445, Paramount, California
  - Site 402, Sacramento, California
  - Site 425, San Diego, California
  - Site 418, Miami, Florida
  - Site 426, Miami, Florida
  - Site 289, Meridian, Idaho
  - Site 390, Augusta, Kansas
  - Site 421, Newton, Kansas
  - Site 422, Wichita, Kansas
  - Site 443, Louisville, Kentucky
  - Site 420, Louisville, Kentucky
  - Site 441, Louisville, Kentucky
  - Site 393, Metairie, Louisiana
  - Site 436, Metairie, Louisiana
  - Site 285, Binghamton, New York
  - Site 429, Asheboro, North Carolina
  - Site 446, Cincinnati, Ohio
  - Site 427, Dayton, Ohio
  - Site 419, Charleston, South Carolina
  - Site 439, Spartanburg, South Carolina
  - Site 308, Bristol, Tennessee
  - Site 444, Kingsport, Tennessee
  - Site 283, Austin, Texas
  - Site 282, Fort Worth, Texas
  - Site 288, San Angelo, Texas
  - Site 395, Layton, Utah
  - Site 431, Salt Lake City, Utah
  - Site 424, Salt Lake City, Utah
  - Site 428, Salt Lake City, Utah
  - Site 440, West Jordan, Utah
  - Site 433, West Jordan, Utah
  - Site 435, West Jordan, Utah
  - Site 438, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Statler VA, Albano FR, Airey J, Sawlwin DC, Graves Jones A, Matassa V, Heijnen E, Edelman J, Marshall GS. Immunogenicity and safety of a quadrivalent inactivated influenza vaccine in children 6-59 months of age: A phase 3, randomized, noninferiority study. Vaccine. 2019 Jan 7;37(2):343-351. doi: 10.1016/j.vaccine.2018.07.036. Epub 2018 Jul 26. PMID 30057283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 27 September 2016 to 11 August 2017 from 39 study sites in the United States of America.
Pre-assignment Details: A total of 2339 subjects were screened. A total of 2250 subjects were randomized to study treatment. Due to not having valid informed consent, 3 subjects were removed from the clinical database. Therefore, overall 2247 subjects gave informed consent and were included in the analysis set.
Groups:
- Seqirus QIV: Subjects 6 months through 59 months of age who received Seqirus Quadrivalent Inactivated Influenza Vaccine.
- Comparator QIV: Subjects 6 months through 59 months of age who received Comparator Quadrivalent Inactivated Influenza Vaccine.
Period: Overall Study
Arm/Group | Seqirus QIV | Comparator QIV
Started ((Randomized)) | 1687 | 563
Included in Clinical Database / FAS | 1684 | 563
Completed | 1566 | 521
Not Completed | 121 | 42
Not completed — Lost to Follow-up | 84 | 29
Not completed — Withdrawal by Subject | 26 | 10
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 3 | 1
Not completed — Other | 4 | 1
Not completed — Excluded due to invalid informed consent | 3 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set was used for analysis of subject characteristics and comprised all subjects whose parent(s)/guardian(s) had given informed consent and who were randomized to treatment. Screening failures were not included in the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Seqirus QIV | Comparator QIV | Total
Number analyzed (Participants) | 1684 | 563 | 2247
Age, Continuous [Mean (Standard Deviation); unit: months] | 36.6 (14.70) | 36.5 (14.68) | 36.6 (14.69)
Age, Customized [Count of Participants; unit: Participants]
  6 through 35 months | 700 | 235 | 935
  36 through 59 months | 984 | 328 | 1312
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 820 | 268 | 1088
  Male | 864 | 295 | 1159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 434 | 160 | 594
  Not Hispanic or Latino | 1243 | 400 | 1643
  Unknown or Not Reported | 7 | 3 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 2 | 7
  Asian | 15 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 13 | 3 | 16
  Black or African American | 361 | 123 | 484
  White | 1205 | 391 | 1596
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 85 | 34 | 119
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1684 | 563 | 2247
Weight [Mean (Standard Deviation); unit: kilograms] | 15.36 (4.224) | 15.40 (4.149) | 15.37 (4.205)
Prevaccination Axillary Temperature [Mean (Standard Deviation); unit: °F] | 97.17 (0.963) | 97.25 (0.935) | 97.19 (0.936)
Vaccination against influenza 2015/2016 season [Count of Participants; unit: Participants] | 845 | 294 | 1139

OUTCOME MEASURES:

1. Primary Outcome: The Geometric Mean Titer (GMT) Ratio of Each Virus Strain.
Description: Noninferiority of Seqirus QIV compared to comparator QIV was assessed by hemagglutination inhibition (HI) antibody geometric mean titer (GMT) for each viral strain included in the vaccines. The GMT ratio is defined as the geometric mean of the postvaccination HI titer for the US-licensed comparator QIV over the geometric mean of the postvaccination HI titer for Seqirus QIV.
  B/VIC = B/Victoria B/YAM = B/Yamagata
Time Frame: Postvaccination (28 days after last vaccination)
Population: The Per-Protocol Population (PPS) comprised all subjects in the Evaluable Population who did not have any protocol deviations that were medically assessed as potentially impacting on immunogenicity results.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Arm/Group | Seqirus QIV | Comparator QIV
Number analyzed (Participants) | 1456 | 484
Geometric Mean Titer
  A/H1N1 | 370.0 [345.13 to 396.55] | 311.7 [276.88 to 350.90]
  A/H3N2: number analyzed (Participants) | 1455 | 484
  A/H3N2 | 436.8 [403.04 to 473.28] | 589.1 [516.42 to 671.91]
  B/YAM | 25.5 [23.93 to 27.06] | 29.7 [26.51 to 33.21]
  B/VIC: number analyzed (Participants) | 1456 | 483
  B/VIC | 56.8 [52.90 to 60.96] | 57.9 [51.04 to 65.62]
Statistical Analysis 1: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to A/H1N1 vaccine strain measured in terms of Geometric Mean Titer ratios 28 days after the last vaccination; Test type: Non-Inferiority — The non-inferiority criterion for the GMT ratio (adjusted analysis) was that the upper bound of the two-sided 95% confidence interval (CI) of the GMT ratio for the Comparator QIV GMT, divided by the Seqirus QIV GMT, should not exceed 1.5; Geometric Mean Titer Ratio = 0.79, 95% CI 2-sided [0.72 to 0.88]
Statistical Analysis 2: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to A/H3N2 vaccine strain measured in terms of Geometric Mean Titer ratios 28 days after the last vaccination; Test type: Non-Inferiority — The non-inferiority criterion for the GMT ratio (adjusted analysis) was that the upper bound of the two-sided 95% CI of the GMT ratio for the Comparator QIV GMT, divided by the Seqirus QIV GMT, should not exceed 1.5; Geometric Mean Titer Ratio = 1.27, 95% CI 2-sided [1.15 to 1.42]
Statistical Analysis 3: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to B/YAM vaccine strain measured in terms of Geometric Mean Titer ratios 28 days after the last vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer Ratio = 1.12, 95% CI 2-sided [1.01 to 1.24]
Statistical Analysis 4: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to B/VIC vaccine strain measured in terms of Geometric Mean Titer ratios 28 days after the last vaccination; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Geometric Mean Titer Ratio = 0.97, 95% CI 2-sided [0.86 to 1.09]

2. Primary Outcome: The Difference in Seroconversion Rate (SCR) for Each Virus Strain.
Description: Noninferiority of Seqirus QIV compared to comparator QIV will be assessed by seroconversion rate (SCR) for each viral strain. SCR is defined as the percentage of subjects with either a prevaccination HI titer < 1:10 and a postvaccination HI titer ≥ 1:40, or a prevaccination HI titer ≥ 1:10 and a ≥ 4-fold increase in postvaccination HI titer. For the SCR comparison, the difference between the SCR for each vaccine (for each strain) will be determined.
Time Frame: Postvaccination (28 days after last vaccination)
Population: The Per-Protocol Population comprised all subjects in the Evaluable Population who did not have any protocol deviations that were medically assessed as potentially impacting on immunogenicity results.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Seqirus QIV | Comparator QIV
Number analyzed (Participants) | 1456 | 484
Percentage of participants
  A/H1N1 | 79.1 [76.9 to 81.1] | 68.8 [64.5 to 72.9]
  A/H3N2: number analyzed (Participants) | 1455 | 484
  A/H3N2 | 82.3 [80.2 to 84.2] | 84.9 [81.4 to 88.0]
  B/YAM | 38.9 [36.4 to 41.4] | 41.9 [37.5 to 46.5]
  B/VIC: number analyzed (Participants) | 1456 | 483
  B/VIC | 60.2 [57.6 to 62.7] | 61.1 [56.6 to 65.4]
Statistical Analysis 1: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to A/H1N1 vaccine strain measured in terms of Seroconversion Rate Difference 28 days after the last vaccination; Test type: Non-Inferiority — The noninferiority criterion for the SCR difference was that the upper bound of the two-sided 95% CI on the difference between SCRs for Comparator QIV minus the Seqirus QIV SCR should not exceed 10%; Seroconversion Rate Difference = -10.3, 95% CI 2-sided [-15.4 to -5.1]
Statistical Analysis 2: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to A/H3N2 vaccine strain measured in terms of Seroconversion Rate Difference 28 days after the last vaccination; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Seroconversion Rate Difference = 2.6, 95% CI 2-sided [-2.54 to 7.8]
Statistical Analysis 3: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to B/YAM vaccine strain measured in terms of Seroconversion Rate Difference 28 days after the last vaccination; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Seroconversion Rate Difference = 3.1, 95% CI 2-sided [-2.1 to 8.2]
Statistical Analysis 4: Comparison: Seqirus QIV vs Comparator QIV; Non-inferiority of immune responses to B/VIC vaccine strain measured in terms of Seroconversion Rate Difference 28 days after the last vaccination; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Seroconversion Rate Difference = 0.9, 95% CI 2-sided [-4.2 to 6.1]

3. Secondary Outcome: Number of Participants With Solicited Local Adverse Reactions and Solicited Systemic Adverse Events (AE)
Description: Frequency and severity of solicited local adverse reactions and systemic AEs for 7 days after each vaccination dose
Time Frame: Postvaccination (up to 7 days after vaccination)
Population: The Solicited Safety Population comprises all subjects in the Full Analysis Set (FAS) who received at least one dose or partial dose of Study Vaccine and had provided any evaluable data on solicited events.
Measure: Count of Participants; unit: Participants
Arm/Group | Seqirus QIV | Comparator QIV
Number analyzed (Participants) | 1618 | 545
Participants
  Solicited AEs, Any | 940 | 312
  Solicited AEs, Grade 1 | 592 | 189
  Solicited AEs, Grade 2 | 277 | 83
  Solicited AEs, Grade 3 | 71 | 39
  Solicited AEs, Local | 645 | 208
  Solicited AEs, Systemic | 633 | 215

4. Secondary Outcome: Number of Participants With Cellulitis-like Reactions
Description: Frequency of cellulitis-like reactions for at least 28 days after each vaccination dose
Time Frame: Postvaccination (up to 28 days after each vaccination)
Population: The Solicited Safety Population comprises all subjects in the FAS who received at least one dose or partial dose of Study Vaccine and had provided any evaluable data on solicited events.
Measure: Count of Participants; unit: Participants
Arm/Group | Seqirus QIV | Comparator QIV
Number analyzed (Participants) | 1618 | 545
Participants | 0 | 1

5. Secondary Outcome: Number of Participants With Unsolicited AEs
Description: Frequency and severity of unsolicited AEs for at least 28 days after each vaccination dose
Time Frame: Postvaccination (up to 28 days after vaccination)
Population: The Overall Safety Population was used for the analysis of overall and unsolicited adverse event safety and comprised all subjects in the FAS who received at least one dose or partial dose of Study Vaccine and have provided any evaluable follow-up safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Seqirus QIV | Comparator QIV
Number analyzed (Participants) | 1673 | 559
Participants
  Unsolicited AEs, Any | 536 | 171
  Unsolicited AEs, Grade 1 | 285 | 92
  Unsolicited AEs, Grade 2 | 206 | 65
  Unsolicited AEs, Grade 3 | 45 | 14

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE)
Description: Frequency of SAEs for 180 days after the last vaccination dose. SAE = serious adverse events, AESI = adverse event of special interest
Time Frame: 180 days after the last vaccination dose.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Seqirus QIV | Comparator QIV
Number analyzed (Participants) | 1673 | 559
Participants
  SAEs (Day 1 to Day 28) | 4 | 0
  SAEs (Day 29 to Final Database Lock) | 7 | 3
  Related SAEs | 0 | 0
  Deaths | 0 | 0
  AESIs (Day 1 to Day 28) | 0 | 0
  AESIs (Day 29 to Final Database Lock) | 2 | 0

7. Secondary Outcome: Geometric Mean of Hemagglutination Titers (HI GMTs) Prevaccination (Day 1) and Postvaccination (Study Exit Visit) of Each Virus Strain
Description: The humoral immune response will be assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains will be used to calculate geometric mean of HI titers prevaccination & postvaccination.
Time Frame: 28 days after last vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Seqirus QIV Cohort A: Subjects 6 months through 35 months of age who received Seqirus Quadrivalent Inactivated Influenza Vaccine.
- Seqirus QIV Cohort B: Subjects 36 months through 59 months of age who received Seqirus Quadrivalent Inactivated Influenza Vaccine.
- Comparator QIV Cohort A: Subjects 6 months through 35 months of age who received Comparator Quadrivalent Inactivated Influenza Vaccine.
- Comparator QIV Cohort B: Subjects 36 months through 59 months of age who received Comparator Quadrivalent Inactivated Influenza Vaccine.
Arm/Group | Seqirus QIV Cohort A | Seqirus QIV Cohort B | Comparator QIV Cohort A | Comparator QIV Cohort B
Number analyzed (Participants) | 586 | 870 | 193 | 291
Titers
  A/H1N1, Prevaccination | 13.8 [12.30 to 15.57] | 60.7 [53.97 to 68.20] | 14.9 [12.25 to 18.22] | 68.7 [55.84 to 84.62]
  A/H1N1, Postvaccination | 184.9 [165.15 to 207.05] | 590.2 [548.62 to 634.93] | 168.3 [137.69 to 205.62] | 469.2 [413.72 to 532.05]
  A/H3N2, Prevaccination | 14.3 [12.48 to 16.39] | 62.4 [55.50 to 70.19] | 16.4 [12.86 to 20.91] | 65.5 [53.76 to 79.88]
  A/H3N2, Postvaccination: number analyzed (Participants) | 585 | 870 | 193 | 291
  A/H3N2, Postvaccination | 184.9 [164.57 to 207.65] | 778.6 [710.83 to 852.82] | 247.5 [202.14 to 302.95] | 1047 [911.69 to 1202.48]
  B/YAM, Prevaccination | 5.9 [5.66 to 6.13] | 7.9 [7.55 to 8.33] | 5.8 [5.47 to 6.22] | 8.3 [7.58 to 9.17]
  B/YAM, Postvaccination | 15.6 [14.33 to 17.00] | 35.4 [32.73 to 38.26] | 16.3 [14.03 to 18.95] | 44.1 [38.30 to 50.87]
  B/VIC, Prevaccination: number analyzed (Participants) | 586 | 870 | 193 | 290
  B/VIC, Prevaccination | 7.1 [6.75 to 7.55] | 9.6 [9.04 to 10.19] | 6.9 [6.26 to 7.53] | 10.4 [9.35 to 11.64]
  B/VIC, Postvaccination | 39.8 [36.02 to 44.04] | 72.1 [65.62 to 79.25] | 31.9 [26.88 to 37.81] | 85.9 [73.16 to 100.96]

8. Secondary Outcome: Seroconversion Rates (SCRs) of Each Virus Strain
Description: The humoral immune response will be assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains will be used to calculate SCRs defined as the % of subjects with either a prevaccination HI titer < 1:10 and a postvaccination HI titer ≥ 1:40 or a prevaccination titer ≥ 1:10 and a ≥ 4-fold increase in postvaccination titer.
Time Frame: 28 days after last vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Seqirus QIV Cohort A | Seqirus QIV Cohort B | Comparator QIV Cohort A | Comparator QIV Cohort B
Number analyzed (Participants) | 586 | 870 | 193 | 291
Percentage of participants
  A/H1N1 | 81.9 [78.6 to 84.9] | 77.1 [74.2 to 79.9] | 80.3 [74.0 to 85.7] | 61.2 [55.3 to 66.8]
  A/H3N2: number analyzed (Participants) | 585 | 870 | 193 | 291
  A/H3N2 | 82.4 [79.1 to 85.4] | 82.2 [79.5 to 84.7] | 85.0 [79.1 to 89.7] | 84.9 [80.2 to 88.8]
  B/YAM | 22.5 [19.2 to 26.1] | 49.9 [46.5 to 53.3] | 26.9 [20.8 to 33.8] | 51.9 [46.0 to 57.8]
  B/VIC: number analyzed (Participants) | 586 | 870 | 193 | 290
  B/VIC | 52.9 [48.8 to 57.0] | 65.1 [61.8 to 68.2] | 49.7 [42.5 to 57.0] | 68.6 [62.9 to 73.9]

9. Secondary Outcome: Seroprotection Rates of Each Virus Strain
Description: The humoral immune response will be assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains will be used to calculate the percentage of subjects with a titer ≥40 (seroprotection rates) at Day 1 and at Study Exit Visit.
Time Frame: 28 days after last vaccination.
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Seqirus QIV Cohort A | Seqirus QIV Cohort B | Comparator QIV Cohort A | Comparator QIV Cohort B
Number analyzed (Participants) | 586 | 870 | 193 | 291
Percentage of participants
  A/H1N1 | 90.1 [87.4 to 92.4] | 99.1 [98.2 to 99.6] | 88.6 [83.3 to 92.7] | 98.3 [96.0 to 99.4]
  A/H3N2: number analyzed (Participants) | 585 | 870 | 193 | 291
  A/H3N2 | 92.5 [90.0 to 94.5] | 98.4 [97.3 to 99.1] | 95.3 [91.3 to 97.8] | 98.6 [96.5 to 99.6]
  B/YAM | 24.7 [21.3 to 28.4] | 57.1 [53.8 to 60.4] | 29.0 [22.7 to 36.0] | 61.5 [55.7 to 67.1]
  B/VIC | 55.6 [51.5 to 59.7] | 71.0 [67.9 to 74.0] | 52.8 [45.6 to 60.1] | 75.3 [69.9 to 80.1]

10. Secondary Outcome: Geometric Mean Fold Increase (GMFI) of Each Virus Strain
Description: The humoral immune response will be assessed for Seqirus QIV & comparator QIV. Serum HI titers against the 4 influenza vaccine strains will be used to calculate GMFIs, defined as the geometric mean fold titer change (rise) from Day 1 to Study Exit Visit.
Time Frame: Prevaccination (Day 1) and Postvaccination (28 days after last vaccination)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | Seqirus QIV Cohort A | Seqirus QIV Cohort B | Comparator QIV Cohort A | Comparator QIV Cohort B
Number analyzed (Participants) | 586 | 870 | 193 | 291
Fold Change
  A/H1N1 | 13.4 [11.98 to 14.90] | 9.7 [8.90 to 10.64] | 11.3 [9.40 to 13.49] | 6.8 [5.83 to 7.99]
  A/H3N2: number analyzed (Participants) | 585 | 870 | 193 | 291
  A/H3N2 | 13.0 [11.62 to 14.50] | 12.5 [11.42 to 13.62] | 15.1 [12.60 to 18.08] | 16.0 [13.62 to 18.74]
  B/YAM | 2.6 [2.45 to 2.86] | 4.5 [4.17 to 4.77] | 2.8 [2.45 to 3.19] | 5.3 [4.67 to 6.00]
  B/VIC: number analyzed (Participants) | 586 | 870 | 193 | 290
  B/VIC | 5.6 [5.11 to 6.09] | 7.5 [6.93 to 8.15] | 4.6 [3.97 to 5.42] | 8.2 [7.18 to 9.42]

ADVERSE EVENTS:
Time Frame: Non-serious unsolicited AEs and serious AEs were collected from Day 1 through Day 180
Description: Of the 2247 subjects who provided consent, 7 subjects discontinued from the study and did not receive any vaccination; and 8 subjects had no reported safety data. Therefore, 2232 subjects were included in the overall safety population.
  Seqirus QIV N = 1673 Comparator QIV N = 559
Arm/Group | Seqirus QIV | Comparator QIV
All-Cause Mortality (participants affected / at risk) | 0/1673 | 0/559
Serious Adverse Events (participants affected / at risk) | 11/1673 | 3/559
Other Adverse Events (participants affected / at risk) | 320/1673 | 80/559
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seqirus QIV (N=1673) | Comparator QIV (N=559)
Croup Infectious (Infections and infestations) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seqirus QIV (N=1673) | Comparator QIV (N=559)
Cough (Respiratory, thoracic and mediastinal disorders) | 153 (167) | 41 (52)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 134 (155) | 53 (63)
Pyrexia (Infections and infestations) | 91 (100) | 25 (29)
Upper respiratory tract infection (Infections and infestations) | 67 (72) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Seqirus agreements and restrictions on publishing may vary with individual investigators; however, Seqirus will not prohibit any investigator from publishing. Seqirus supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT02914275/Prot_000.pdf
  • Statistical Analysis Plan (2016-08-22): https://cdn.clinicaltrials.gov/large-docs/75/NCT02914275/SAP_001.pdf